CLINICAL TRIAL: NCT04925960
Title: A Prospective, Randomized, Double-Blind, Placebo-Controlled, Single-Center Study of Oral Epalrestat Therapy in Pediatric Subjects With Phosphomannomutase 2-congenital Disorder of Glycosylation (PMM2-CDG)
Brief Title: Oral Epalrestat Therapy in Pediatric Subjects With PMM2-CDG
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to futility
Sponsor: Maggie's Pearl, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 21-000492
Record Dates: First submitted 2021-06-08; First posted 2021-06-14 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Pmm2-CDG; Phosphomannomutase 2 Deficiency; Phosphomannomutase 2 Congenital Disorder of Glycosylation; Phosphomannomutase II Congenital Disorder of Glycosylation; Phosphomannomutase II Deficiency
MeSH Terms: conditions — Congenital disorder of glycosylation type 1A | interventions — epalrestat

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to treatment or placebo. Patients and study staff will be blinded to the study arm.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients and all study personnel will remain blinded to the original treatment assignment until study close.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Epalrestat (Experimental): Epalrestat will be administered orally, 3 times per day (TID) spaced out as evenly as possible over 24 hours in a divided dose starting on Day 1 of the Study.
  Interventions: Drug: Epalrestat
- Placebo (Placebo Comparator): Placebo will be administered orally, 3 times per day (TID) spaced out as evenly as possible over 24 hours in a divided dose starting on Day 1 of the Study.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Epalrestat — Epalrestat is a noncompetitive and reversible aldose reductase inhibitor (ARI) used for the treatment of diabetic neuropathy in Japan. The drug's ability to safely improve symptoms of neuropathy alone by reducing oxidative stress, increasing glutathione levels, and reducing intracellular sorbitol accumulation make it a desirable medication for PMM2-CDG patients who commonly suffer with various neuropathies. However, work recently conducted by Perlara, a public benefit company with the mandate to screen existing commercially available drugs for possible application in rare diseases, has demonstrated that Epalrestat can also elevate the level PMM2 produced endogenously. This may reduce the severity of the morbidities associated with PMM2-CDG.
  Arms: Epalrestat
Drug: Placebo — The placebo capsule with be identical in appearance to the Epalrestat capsule. It will contain microcrystalline cellulose filler in a gelatin capsule.
  Arms: Placebo

SUMMARY:
This is a prospective, single-center, randomized, double-blind, placebo-controlled study designed to assess the safety, tolerability, and clinical and metabolic improvement of pediatric subjects with PMM2-CDG on oral epalrestat therapy vs. placebo.

DETAILED DESCRIPTION:
This is a prospective, single-center, randomized, double-blind, placebo-controlled study designed to assess the safety, tolerability, and clinical and metabolic improvement of pediatric subjects with PMM2-CDG on oral epalrestat therapy vs. placebo. The primary study objective is to evaluate the safety and probable benefit of oral epalrestat therapy in pediatric subjects with PMM2-CDG. Study outcomes include evaluating the metabolic improvement of pediatric subjects treated with oral epalrestat therapy compared to placebo, evaluating safety, clinical improvement, and pharmocokinetics (PK) of oral epalrestat therapy in pediatric subjects compared to placebo, and evaluating urine polyols, adverse events, laboratory data, other safety measures, PK, and Quality of Life surveys to measure clinical improvement.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 2 and < 18 years
2. Diagnosis of PMM2-CDG, based on molecularly confirmed biallelic PMM2 pathogenic variants (can be historical diagnosis with lab report on file)
3. Informed consent (and assent, as applicable) document personally signed by the legally authorized representative of the patient, indicating that the patient's parent/guardian has been informed and agreed to all aspects of the study
4. Be willing and able to adhere to the study assessments and schedule described in the protocol and consent/assent documents
5. Negative urine pregnancy test (only for female subjects of child-bearing potential)
6. For subjects of child-bearing potential-only, subject has been counseled on and agrees to the requirement either for double barrier contraceptive methods and/or for total abstinence from prior to randomization through 3-months after the cessation of treatment.

Exclusion Criteria:

1. Known or suspected other known CDG
2. Known allergy to aldose reductase inhibitors
3. Hypersensitivity to epalrestat
4. Hepatic impairment defined as any one of the following:

   1. AST/ALT >5x ULN in the 6 months prior to screening
   2. Bilirubin >2X ULN in the last 6 months prior to screening
   3. Synthetic liver dysfunction (albumin deficiency < 2.8 mmol/L) at screening, or
   4. Diagnosis of liver fibrosis (Fibroscan > 7 kPa) confirmed by liver elastogram at screening
5. Renal impairment defined as serum creatinine: > 0.5 mg/dL (≤ 6 years); > 0.7 mg/dL (7-10 years); > 1.24 mg/dL (≥ 11 years)
6. Low platelet count (< 125x109 /L)
7. Any other clinically significant lab abnormality which, in the opinion of the investigator, should be exclusionary
8. Anemia (Hgb < 10 g/dL)
9. Use of an investigational drug, including acetazolamide, in the past 28 days; use of an investigational biologic in the past 12 months
10. Concurrent or planned participation in interventional protocol or use of any other unapproved therapeutics, and,
11. Any other medical condition, which, in the opinion of the investigator, will interfere with the patient's ability to comply with the protocol, compromises patient safety, or interferes with the interpretation of the study results.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2022-11-10 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Change in sorbitol (mmol/mol creatinine) | 9 months
  Change in sorbitol from baseline between study arms
Change in ICARS | 9 months
  Change in ICARS from baseline between study arms
Change in Antithrombin III (ATIII) | 9 months
  Change in ATIII from baseline between study arms

SECONDARY OUTCOMES:
Change of Body Max Index (BMI) percentile | 9 months
  Change of BMI percentile from baseline between study arms
Change of factor XI activity percentage | 9 months
  Change of factor XI activity from baseline between study arms
Change of liver transaminases (U/L) | 9 months
  Change of liver transaminases from baseline between study arms
Change of transferrin glycosylation (ratio) | 9 months
  Change of transferrin glycosylationfrom baseline between study arms
Change in Nijmegen Pediatric CDG Rating Scale (NPCRS) score | 9 months
  Change in NPCRS from baseline between study arms
Change of normalized mannitol (mmol/mol creatinine) | 9 months
  Change of normalized mannitol from baseline between study arms

CONTACTS AND LOCATIONS:
Overall Officials: Eva Morava-Kozicz, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided